CLINICAL TRIAL: NCT03488550
Title: A Phase 1, Open-label, Single-dose, Dose-escalation, Safety, Tolerability, and PK Study of Intravitreal ANX007 in Participants With Primary Open-angle Glaucoma
Brief Title: Single-dose Study of ANX007 in Participants With Primary Open-angle Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANX007-GLA-01
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ANX007-GLA-01 (Experimental)
  Interventions: Biological: ANX007

INTERVENTIONS:
Biological: ANX007 — Single ascending dose

SUMMARY:
This is a multi center, open-label, single dose, safety study. Approximately 9 to 15 participants with open-angle glaucoma are assigned into 3 sequential dose-levels and will receive ANX007 administered as single, IVT injections.

DETAILED DESCRIPTION:
This is a phase 1, open-label, dose-escalation, safety study evaluating up to 3 dose levels of ANX007 administered as single IVT injections. Approximately 9 to 15 eligible participants are enrolled into one cohort each. All participants receive ANX007 in an open-label manner. The primary objective is to evaluate the safety and tolerability of a single intravitreal (IVT) injection of ANX007 in participants with primary open-angle glaucoma. Secondary objectives are to evaluate the serum pharmacokinetics (PK) and immunogenicity. An exploratory objective will evaluate the pharmacodynamic (PD) effect of ANX007 on serum C1q activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 years and older
* Diagnosis of primary open-angle glaucoma
* Intraocular pressure <21 mm Hg on a stable IOP treatment regimen
* Reliable visual field testing

Exclusion Criteria:

* BCVA worse than 20/80 in either eye
* Extensive glaucomatous visual-field damage
* History of intraocular inflammatory or infectious eye disease in study eye
* Ocular trauma in study eye within the preceding 6 months
* History of uncomplicated cataract surgery less than 6 mos prior
* Any abnormality preventing reliable Tonopen tonometry in study eye
* Active malignancy within past 5 yrs
* Previous tx with another humanized monoclonal antibody
* History of any autoimmune or neurologic disease
* Concurrent use of glucocorticoid medications
* Receiving monoamine oxidase inhibitor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by the occurrence of adverse events | Day 56

SECONDARY OUTCOMES:
Serum plasma concentration of ANX007 after a single IVT injection. | Day 15
Immunogenicity of ANX007 after a single IVT injection. | Day 56

OTHER OUTCOMES:
Effect of a single IVT injection of ANX007 on serum C1q | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Eric Humphriss, Study Director — Annexon Vice President of Clinical Operations
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

REFERENCES:
- See also: Related Info — http://www.annexonbio.com